CLINICAL TRIAL: NCT03393988
Title: A Pilot Study for a Prospective, Randomized Controlled Trial of Techniques for Perioperative Analgesia for Live Liver Donors
Brief Title: Techniques for Perioperative Analgesia for Live Liver Donors; A Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rasha Samir Abd-ElWahab Bondok, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R45/2017
Record Dates: First submitted 2017-12-23; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia
Keywords: Transversus abdominis plane block,; Dexmedetomidine; Fentanyl; Live liver donor; Liver transplantation
MeSH Terms: interventions — Analgesics, Opioid; Anesthesia, Conduction; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group F (Active Comparator): Fentanyl infusion (0.5 µg/kg/hr)
  Interventions: Drug: Fentanyl infusion
- Group (TAP-Dex) (Active Comparator): Ultrasound guided TAP block and Dexmedetomidine
  * Ultrasound guided subcostal oblique TAP block with 0.25 % bupivacaine
  * Dexmedetomidine infusion(200 µg in 2 ml diluted in 48 ml of saline)
  * Fentanyl infusion (0.5 µg/kg/hr).
  Interventions: Drug: Fentanyl infusion; Procedure: Ultrasound guided TAP block; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl infusion — After induction of general anesthesia; Fentanyl infusion (0.5 µg/kg/hr) will be started (which will be afterwards adjusted intraoperatively according to the hemodynamics and Bispectral Index (BIS) reading).
  Other Names: Opioid
Procedure: Ultrasound guided TAP block — After induction of general anesthesia; Patients will receive ultrasound guided subcostal oblique TAP block with 0.25 % bupivacaine 40 ml on each side resulting in a total volume of 80 ml, subcostal TAP block was given twice, at the beginning and at the end of the surgery.
  Other Names: Regional anesthesia
  Arms: Group (TAP-Dex)
Drug: Dexmedetomidine — Dexmedetomidine (200 µg in 2 ml diluted in 48 ml of saline) will be started in a dose of 1 μg/kg over 10 min then maintenance dose as continuous infusion between 0.2 and 0.8 μg/ kg/h through infusion pump (which will be adjusted according to the hemodynamics and BIS reading)
  Other Names: alpha 2 sympathomimetic
  Arms: Group (TAP-Dex)

SUMMARY:
This study,will evaluate the efficacy of ultrasound (US)-guided subcostal oblique TAP block together with IV infusion of Dexmedetomidine and fentanyl as a type of multimodal analgesic regimen in comparison with IV fentanyl based analgesia only in live liver donors.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) physical status I or II
* Scheduled as live liver donors
* J-shaped incision in the supraumblical region

Exclusion Criteria:

* Patients with a history of psychiatric/neurological illness,
* Hypertensive patients,
* Morbidly obese patients,
* Pregnant and nursing women,
* Patients with known allergic reaction to any of the study medications,
* Patients on recent use of sedatives or analgesics,
* Patients with significant laboratory abnormalities

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Total fentanyl consumption | Intraoperative
  Total Intravenous fentanyl consumption during the operation

SECONDARY OUTCOMES:
Average sevoflurane concentration | Intraoperative
  The average sevoflurane concentration (the average concentration (%) for the case will be determined from the vaporizer setting recorded in the anesthetic record per 5-minute interval)
The severity of postoperative nausea and vomiting (PONV) | First 24 hours postoperatively
  Will be recorded and classified as "no PONV, mild PONV, moderate PONV and severe PONV"
Ramsay sedation score (RSS) | First 24 hours postoperatively
  Will be used for assessment of sedation immediately after extubation, after 2 hours of ICU admission, after 12 hours then after 24 hours .

CONTACTS AND LOCATIONS:
Locations (1):
- Hospitals of Faculty of Medicine , Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided